CLINICAL TRIAL: NCT07259213
Title: A Phase 1/2a Study to Evaluate the Safety, Tolerability, Whole-Body Distribution, and Preliminary Clinical Activity of 161Tb-RAD402, a Radiolabeled Anti-Kallikrein-Related Peptidase 3 (KLK3) Monoclonal Antibody Targeting Free Prostate-Specific Antigen, in Participants With Castration-Resistant Prostate Cancer (CRPC)
Brief Title: A Study of Terbium 161 (161Tb)-RAD402 in Participants With CRPC
Acronym: RAD402
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Radiopharm Theranostics, Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RAD402-AU-101
Record Dates: First submitted 2025-11-15; First posted 2025-12-02 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Castration-resistant Prostate Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- 161Tb RAD402 (Experimental): Single-arm, open-label study of 161Tb RAD402 consisting of Phase 1 Dose Escalation and Phase 2 Dose Expansion study parts.
  Interventions: Drug: 161Tb RAD402

INTERVENTIONS:
Drug: 161Tb RAD402 — 161Tb RAD402 administered at treatment doses

SUMMARY:
A Phase 1/2a Study to Evaluate the Safety, Tolerability, Whole-Body Distribution, and Preliminary Clinical Activity of 161Tb-RAD402, a Radiolabeled Anti-KLK3 Monoclonal Antibody Targeting Free Prostate-Specific Antigen, in Participants with Castration-Resistant Prostate Cancer (CRPC).

DETAILED DESCRIPTION:
The purpose of this study is to establish the safety profile, biodistribution, pharmacokinetics (PK), and radiation dosimetry of 161Tb-RAD402, to determine the maximum tolerated dose (MTD) and/or recommended Phase 2 dose (RP2D), and to evaluate preliminary anti-tumor activity in participants with locally advanced or metastatic Castration-Resistant Prostate Cancer (CRPC).

The study is divided into 2 phases. Phase 1 is the dose escalation phase to establish the safety profile of 161Tb-RAD402 and to determine the MTD and/or RP2D of 161Tb-RAD402 using a Bayesian Optimal Interval (BOIN) design. Phase 2a is the dose expansion phase at the RP2D to confirm the safety of the MTD and/or RP2D and to evaluate preliminary anti-tumor activity of 161Tb-RAD402 using a probability of success design for Prostate Specific Antigen (PSA)50 based on a Bayesian beta-binomial design.

Participants ≥ 18 years of age with CRPC who have documented disease progression during or after their most recent line of anticancer therapy will be eligible to enroll.

Each phase consists of a Screening Period, a Treatment and Imaging Period, and a Safety and Long-term Follow-up Period.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide informed consent prior to start of any study procedures and assessments and must be willing to comply with all study procedures.
* Male participants ≥ 18 years of age.
* Participants with a documented history of histopathologically confirmed locally advanced or metastatic CRPC defined as follows:

  1. Progressive CRPC defined as castrate levels of testosterone and progressing by at least one of the following criteria:

     * Serum PSA increase >25% and >2.0 ng/ml above nadir, confirmed by progression at 2 timepoints at least 3 weeks apart (PCWG3)
     * Soft tissue progression defined as a ≥20% increase in the sum of the diameter (short axis for nodal lesions and long axis for non-nodal lesions) of all target lesions based on the smallest sum of the diameter since the previous treatment was started or the appearance of one or more new lesions by computed tomography (CT)/ magnetic resonance imaging (MRI).
     * Progression of bone disease defined by PCWG3 as evaluable disease or new bone lesions by bone scan (if metastatic disease).
     * Identification of new soft tissue or bone lesions on PSMA PET imaging.
  2. If metastatic disease, metastatic disease defined as either or both of the following:

     * Documented M1 disease on conventional imaging (CT/MRI of the chest/abdomen/pelvis and/or Technetium 99m [99mTc] whole-body bone scan)
     * Identification of bone lesion(s), extra-pelvic soft tissue lesion(s), or visceral metastases on PSMA PET imaging with an FDA-approved imaging agent (e.g., Gallium-68 (68Ga)-PSMA-11)
  3. PSMA PET-positive disease, defined as at least one PSMA-positive metastatic lesion PSMA PET-positive lesions are defined as uptake greater than that of liver parenchyma in one or more extra-pelvic metastatic lesions of any size in any organ system using an FDA-approved PSMA PET imaging agent.
  4. Progression following treatment with androgen deprivation therapy (ADT) and at least one androgen receptor signaling inhibitor (ARSI) (e.g., enzalutamide, apalutamide, darolutamide, and/or abiraterone acetate). If a participant is currently on ADT, they should continue ADT for the duration of their participation in the study but will not be permitted to start a new therapy or ADT regimen. If a participant has progressed on an ARSI, they will have the option to remain on the same ARSI or discontinue therapy.
  5. Prior definitive and palliative external beam radiation therapy and stereotactic body radiation therapy is allowed.

Note: Participants with extended external beam radiation therapy to the axial skeleton, which in the opinion of the Investigator may pose a risk for increased myelotoxicity, will be discussed with the Sponsor to determine eligibility.

* Prior treatment with lutetium (Lu-177)-PSMA-radioligand (RL), defined as up to 6 doses of lutetium (177Lu) vipivotide tetraxetan (Pluvicto) or investigational use of up to 4 doses of Lu-177-PSMA-imaging and treatment (I&T) is allowed but not required.

  a. Prior treatment with (no more than) one taxane-based chemotherapy is allowed but not required. A taxane-based chemotherapy is defined as a minimum exposure of two cycles of a taxane chemotherapy.
* Participants must have documented disease progression during or after their most recent line of anticancer therapy.
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1.
* Participants must have a life expectancy of ≥ 4 months in the opinion of the Investigator.
* Participants who are able to father a child must agree to avoid impregnating a partner and to adhere to a highly effective method of contraception during the study and for 6 months after the last dose of 161Tb-RAD402. All participants must agree to not donate sperm during the study and for 6 months after the last dose of 161Tb-RAD402.
* Participants with previously treated brain metastases are eligible to participate if:

  1. they are neurologically and radiologically stable (no evidence of progression by imaging; same imaging modality (MRI or CT scan) must be used for each assessment) for at least 28 days prior to the first dose of 161Tb-RAD402; and
  2. do not require corticosteroids at a dose of >10 mg prednisolone equivalent to treat associated neurological symptoms, and
  3. have no history of leptomeningeal disease or spinal cord compression.

Exclusion Criteria:

* Prostate cancer with known significant sarcomatoid, or spindle cell, or neuroendocrine small cell components, or metastasis of other cancer to the prostate.
* History of prior organ transplant (other than corneal transplant)
* Any other known, active malignancy except for non-melanoma skin cancer or adequately treated non-muscle-invasive urothelial carcinoma of the bladder (i.e. tumor in situ (Tis), tumor grade a (Ta) and low-grade tumor grade 1 (T1) tumors). Participants with a history of malignancies of low recurrence potential who have received curative-intent therapy may be approved on a case-by-case basis in discussion with the Sponsor, if it is determined not to put the participant at an increased risk of adverse drug effects and/or interfere with the integrity of the study outcome.
* Have any medical condition that would, in the Investigator's judgment, prevent the participant's full participation in the clinical study due to safety concerns or compliance with clinical study procedures such as participants with severe claustrophobia who are unresponsive to oral anxiolytics, participants with low back pain who cannot lie comfortably on an imaging table, participants who are hyperactive or hyperkinetic such that they cannot tolerate lying still for multiple time point imaging procedures, etc.
* Residual toxicity ≥ Grade 2 from prior anti-cancer therapy (except alopecia and peripheral sensory neuropathy).
* History of uncontrolled allergic reactions and/or known or expected hypersensitivity to protein therapeutics, 161Tb-RAD402, or any of its excipients.
* Inadequate organ functions as reflected in laboratory parameters:

  * Estimated glomerular filtration rate (eGFR) < 50 mL/min adjusted for body surface area (BSA) using the Chronic Kidney Disease Epidemiology Collaboration formula
  * Platelet count of < 100 x 109/L
  * Absolute neutrophil count (ANC) < 1.5 x 109/L
  * Hemoglobin < 9 g/dL
  * Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 3 x upper limit of normal (ULN), or > 5 x ULN for participants with known liver metastases
  * Total bilirubin > 1.5 x ULN, except for participants with documented Gilbert's syndrome who are eligible if total bilirubin ≤ 3 x ULN
  * For participants not taking warfarin or other anticoagulants: International Normalised Ratio (INR) ≤1.5 or PT ≤1.5 x ULN; and either partial thromboplastin time or activated partial thromboplastin time (PTT or aPTT) ≤1.5 x ULN. Participants taking warfarin must be on a stable dose that results in a stable INR <3.5. Among participants receiving other anticoagulant therapy, PT or aPTT must be within the intended therapeutic range of the anticoagulant.
* Participants requiring blood product transfusion within 2 weeks of first dose of 161Tb-RAD402 are not eligible to participate.
* Clinically significant cardiovascular disease including but not limited to:

  * Unstable angina
  * Acute myocardial infarction within 6 months prior to screening
  * New York Heart Association (NYHA) Class II or greater congestive heart failure
  * Clinically significant abnormalities in rhythm, conduction or morphology on resting electrocardiogram (ECG) (e.g., complete left bundle branch block, third degree heart block)
  * Known left ventricular ejection fraction (LVEF) < 50%
  * QT corrected using Fridericia's formula (QTcF) > 480 msec on screening ECG, or congenital long QT syndrome.
* Participation in any other interventional investigational trial for treatment of the underlying malignancy at the time of informed consent signature.
* Major surgery within 4 weeks prior to first dose of 161Tb-RAD402.
* Received prior therapy with a poly (ADP-ribose) polymerase (PARP) inhibitor or radium Ra 223 dichloride (Xofigo). Prior treatment with Lu-177-PSMA-radioligand (RL) is allowed.
* Received anti-cancer therapy, including chemotherapy, immunotherapy, radiation therapy, biologic, herbal therapy, or any investigational therapy or investigational device, within 28 days (or 5 half-lives for biologic/non-cytotoxic agents, whichever is shorter), prior to the first dose of 161Tb-RAD402. For participants who received radiotherapy more than 28 days prior to the first dose of 161Tb-RAD402, efforts should be made to calculate the prior radiation absorbed dose to each critical organ such as the kidneys, liver, lungs, and bone marrow.
* Known active hepatitis B (defined as hepatitis B surface antigen [HBsAg] reactive) or known active hepatitis C virus (HCV) (defined as HCV ribonucleic acid (RNA) [qualitative] is detected) infection. Active viral (any etiology) hepatitis participants are excluded. Participants with serologic evidence of chronic hepatitis B virus (HBV) infection (defined by a positive hepatitis B surface antigen test and a positive anti hepatitis core antigen antibody test) who have a viral load below the limit quantification (HBV deoxy ribonucleic acid (DNA) titer < 1000 copies/mL or 200 international units (IU)/mL) and are not currently on viral suppressive therapy may be eligible and should be discussed with the Sponsor's Medical Monitor (or designee). Note, participants with a history of HCV infection should have completed curative antiviral treatment and have a viral load below the limit of quantification to be eligible to enroll into the study. No testing for HBV or HCV is required unless mandated by local health authority.
* Any uncontrolled intercurrent illness or clinically significant uncontrolled condition(s), including but not limited to active bacterial, fungal, or viral infections requiring systemic therapy.
* Untreated moderate to severe hydronephrosis. If hydronephrosis is corrected via stent or nephrostomy, hydronephrosis will be considered resolved.
* Superscans by nuclear medicine/99mTc bone scan.
* Active autoimmune disease that has required systemic treatment within 90 days (i.e., with the use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid [stable / low doses of ≤10 mg/day prednisone or equivalent dose]) for adrenal or pituitary insufficiency is not considered a form of systemic treatment and is allowed.
* Any other clinically significant comorbidities, such as uncontrolled pulmonary disease, active infection, or any other condition (e.g., prior organ transplant), which in the judgment of the investigator could compromise compliance with the protocol, interfere with the interpretation of study results, or predispose the subject to safety risks.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Individuals' gender of male physical characteristics is the primary criterion for inclusion.
Enrollment: 73 (Estimated)
Dates: Start 2026-02-20 (Estimated); Primary Completion 2028-11-30 (Estimated); Study Completion 2029-03-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment emergent adverse events of 161Tb RAD402 (phase 1) (Safety) | 6 weeks
  As defined per Common Terminology Criteria for Adverse Events (CTCAE) v5.0
Recommended dose(s) of 161Tb RAD402 for future exploration (phase 1) | 6 weeks
  Incidence of dose-limiting toxicities (DLTs) during the first 6 weeks following the first 161Tb RAD402 injection
Preliminary anti-tumor activity, as defined by biochemical response, in participants who are treated with 161Tb RAD402 at the RP2D (phase 2a) | Up to 30 weeks
  Proportion of participants who achieve a ≥50% decline in prostate-specific antigen (PSA) 50

SECONDARY OUTCOMES:
Preliminary anti-tumor activity of 161Tb RAD402 (phase 1) | Up to 30 weeks
  As assessed by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1
Preliminary anti-tumor activity of 161Tb RAD402 as defined by biochemical response (phase 1) | Up to 30 weeks
  Proportion of participants who achieve a ≥50% decline in prostate-specific antigen (PSA) 50
Pharmacokinetics of 161Tb RAD402 (phase 1) | 120 hours
  Half-life of 161Tb RAD402 in blood
Radiation dosimetry of 161Tb RAD402 (phase 1) | 120 hours
  Absorbed radiation doses of 161Tb RAD402 in critical organs (e.g., kidneys, bone marrow)
Biodistribution of 161Tb RAD402 (phase 1) | 120 hours
  Time-integrated activity coefficients of 161Tb RAD402 in organs and tumor lesions
Preliminary anti-tumor activity of 161TbRAD402 at the RP2D in participants with Prostate Specific Membrane Antigen (PSMA) Positron Emission Tomography (PET) positive CRPC previously treated with ≥1 Androgen Receptor Signalling Inhibitor (ARSI) (phase 2a) | Up to 30 weeks
  As assessed by Prostate Cancer Working Group (PCWG) 3
Incidence of treatment emergent adverse events of 161Tb RAD402 at the RP2D (phase 2a) (safety and tolerability) | 6 weeks
  As defined per Common Terminology Criteria for Adverse Events (CTCAE) v5.0
Pharmacokinetics of 161Tb RAD402 at the RP2D (phase 2a) | 120 hours
  Half-life of 161Tb RAD402 in blood
Radiation dosimetry of 161Tb RAD402 at the RP2D (phase 2a) | 120 hours
  Absorbed radiation doses of 161Tb RAD402 in critical organs (e.g., kidneys, bone marrow)
Biodistribution of 161Tb RAD402 at the RP2D (phase 2a) | 120 hours
  Time-integrated activity coefficients of 161Tb RAD402 in organs and tumor lesions
Preliminary anti-tumor activity, of 161Tb RAD402 at the RP2D in participants with PSMA PET-positive CRPC who were previously treated with at least one ARSI by comparing the Radiographic progression free survival (rPFS) (phase 2a) | Up to 30 weeks
  As assessed by disease response using RECIST v1.1

IPD SHARING:
Plan to Share IPD: No